CLINICAL TRIAL: NCT04450810
Title: Evaluation of Serum and Salivary NLRP3 in Periodontitis and Diabetes Patients
Brief Title: Role of NLRP3 in Periodontitis and Diabetes
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Researcher, University of Messina
Other Study IDs: 23-18
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Metabolic Disease; Periodontal Diseases
MeSH Terms: conditions — Metabolic Diseases; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Evaluation of serum and salivary NLRP3
  Interventions: Other: Observation of serum and salivary NLRP3 levels
- Periodontitis: Evaluation of serum and salivary NLRP3
  Interventions: Other: Observation of serum and salivary NLRP3 levels
- Diabetes: Evaluation of serum and salivary NLRP3
  Interventions: Other: Observation of serum and salivary NLRP3 levels
- Periodontitis + diabetes: Evaluation of serum and salivary NLRP3
  Interventions: Other: Observation of serum and salivary NLRP3 levels

INTERVENTIONS:
Other: Observation of serum and salivary NLRP3 levels — Evaluation of serum and salivary NLRP3 levels

SUMMARY:
NLRP3 plays a key role in endothelial function and may be a link for the known interaction of periodontitis and diabetes. The investigators compared the impact of gingival health, periodontitis (CP), diabetes or of both diseases (CP +diabetes) on saliva and serum NLRP3levels.

DETAILED DESCRIPTION:
The aim of this study was to evaluate a possible association between NLRP3 and gingival health, periodontitis (CP), diabetes or of both diseases (CP +diabetes) on saliva and serum NLRP3 levels.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 15 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy controls (n=32), periodontitis (n=34), diabetes (n=33), and a combination of periodontitis + diabetes (n=34)
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | 1-year
  evaluation of changes in clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matarese, Study Chair — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: 10 tears
Access Criteria: pubmed